CLINICAL TRIAL: NCT02247908
Title: A Randomized Controlled Trial Evaluating the Impact of Graphic Cigarette Warnings on Smoking Behavior
Brief Title: Impact of Graphic Cigarette Warnings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-2861; 3P30CA016086-38S2 (NIH)
Record Dates: First submitted 2014-09-09; First posted 2014-09-25 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Smoking
Keywords: Cigarette smoking; Smoke; Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Cigarette Smoking; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Graphic Warning (Experimental): Graphic warnings that include text and an image depicting a health effect of smoking will be applied on labels that cover the top half of the front and back of participants' cigarette packs each week for 4 weeks. Within the graphic warning condition, participants will be assigned to receive 1 of 4 warnings for 4 weeks. The text for these warnings was selected from the 2009 Family Smoking Prevention and Tobacco Control Act and the images were proposed by the FDA.
  Interventions: Other: Graphic Warning
- Surgeon General's Warning (Active Comparator): Labels with Surgeon General's Warning text will be applied to the side of participants' cigarette packs each week for 4 weeks, on top of the Surgeon General's Warning printed by the manufacturer.
  Interventions: Other: Surgeon General's Warning

INTERVENTIONS:
Other: Surgeon General's Warning — Participants will be randomly assigned to receive warnings with one of the four Surgeon General's Warnings on their cigarette packs for 4 weeks:
  1. SURGEON GENERAL'S WARNING: Smoking Causes Lung Cancer, Heart Disease, Emphysema, and May Complicate Pregnancy.
  2. SURGEON GENERAL'S WARNING: Quitting Smoking Now Greatly Reduces Serious Risks to Your Health.
  3. SURGEON GENERAL'S WARNING: Smoking by Pregnant Women May Result in Fetal Injury, Premature Birth, and Low Birth Weight.
  4. SURGEON GENERAL'S WARNING: Cigarette Smoke Contains Carbon Monoxide.
  Arms: Surgeon General's Warning
Other: Graphic Warning — Participants will be randomly assigned to receive one of the following four graphic warnings on their cigarette packs for 4 weeks:
  1. Text: "WARNING: Cigarettes are addictive." Image: Man smoking through tracheotomy hole.
  2. Text: "WARNING: Cigarettes causes fatal lung disease." Image: Healthy lungs next to diseased lungs.
  3. Text: "WARNING: Cigarettes cause cancer." Image: Mouth with cancerous lesion on lip.
  4. Text: "WARNING: Smoking can kill you." Image: Woman dying from cancer.
  Arms: Graphic Warning

SUMMARY:
The purpose of this randomized controlled trial is to determine whether graphic health warnings on cigarette packs are more effective than the existing Surgeon General's warning on cigarette packs at encouraging quit attempts. While previous experiments evaluating candidate graphic warnings have been informative, they have used psychological outcomes, such as attitudes or quit intentions, but not actual cessation behavior (e.g., quit attempts). Furthermore, they typically expose participants to warnings in controlled but artificial experimental settings for a short period of time, using much lower frequency and shorter duration of warning exposure than found in the real world. This study addresses these issues by evaluating the impact of warnings on quit attempts by randomly assigning smokers to have their cigarette packs labeled with either a graphic warning or a Surgeon General's warning for four weeks.

Main hypothesis: Smokers randomized to receive graphic warnings on their cigarette packs will be more likely to report a quit attempt in the 4 weeks of the study than smokers randomized to receive a Surgeon General's label on their cigarette packs.

Secondary hypothesis: Smokers randomized to receive graphic warnings on their cigarette packs will have higher quit intentions at 4 weeks than smokers randomized to receive a Surgeon General's label on their cigarette packs, controlling for baseline quit intentions.

DETAILED DESCRIPTION:
The U.S. Food and Drug Administration (FDA) proposed 9 new graphic warnings for cigarette packs in June 2011 to comply with the Family Smoking Prevention and Tobacco Control Act. However, tobacco industry litigation has delayed implementation of graphic warnings. A court ruling that struck down the labels criticized FDA for failing to "present any data - much less the substantial evidence required under the federal law - showing that enacting their proposed graphic warnings will accomplish the agency's stated objective of reducing smoking rates." This study will address this critique head-on by rigorously testing the impact of the graphic warnings on quit attempts in a randomized control trial.

Recruitment: Smokers will first undergo screening online or call the study center to complete the screening questionnaire over the phone. Study staff will schedule eligible smokers for 5 in-person visits. For each of their first 4 visits, smokers will be asked to bring the number of cigarettes they expect to smoke in an 8 day period.

Informed Consent: Prior to consenting smokers, research staff will visually inspect photo identification of smokers who report or appear to be under age 27. At the beginning of the first appointment, study personnel will explain the consent form and ask the smoker to read the form. Once the participant has finished reading the form, the study personnel member will ask the participant if he or she has any questions. Then both parties will sign the consent form and the participant will receive a copy of the consent form.

Randomization: After smokers have consented to participating in the study, study personnel will randomly assign them to a condition. The investigators will determine the randomization order a priori. Smokers have an equal chance of being randomized to receive one of four graphic warnings or one of four Surgeon General's warnings. They will receive the same warning on their packs during the study.

Assessment: Participants will complete 6 computer-based surveys during the study. The first appointment will take around 60 minutes and each subsequent visit will take around 30-45 minutes to complete. At their first visit, they will complete a "baseline pre-test," after which study personnel will show participants one of their cigarette packs with the assigned warning. Participants will be allowed to examine the pack. They will then return the pack to the study personnel and complete a "baseline post-test." At the next 3 appointments, participants will complete only one survey and their packs will be labeled. At the final appointment, they will only complete a survey.

Detailed description of the intervention: While participants are taking the survey, research staff will apply study warning labels to participants' cigarette packs during the first 4 visits. Participants assigned to the graphic warning condition will receive one of four graphic warning labels that will be applied and cover the top half of the front and back of their cigarette packs. The text for the graphic warnings was selected from the 2009 Family Smoking Prevention and Tobacco Control Act and the images were proposed by the FDA. Participants in the Surgeon General's warning condition will receive one of four Surgeon General's Warnings that will be placed on the side of their packs on top of the Surgeon General's warning printed by the manufacturer. This procedure for the control condition is intended to control for the effects of labeling. The investigators will instruct participants in both conditions to use cigarettes from these labeled packs while they are in the study. Each week they will bring in 8 days' of cigarettes (one extra day to provide a buffer in case of rescheduled appointments or smoking more than anticipated) for labeling. Additionally, they will bring in any unused labeled packs from the previous appointment. The investigators will assess how many cigarettes participants smoke from labeled (i.e., study) and unlabeled (i.e., non-study) packs to calculate intervention dose (% of cigarettes smoked from labeled packs). At the end of the study, participants will receive a list of cessation resources. During the final appointment, participants will also report whether they knew anyone else in the study or saw another participant's labels, to assess potential contamination.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Have smoked at least 100 cigarettes in his or her lifetime
* Currently smoke cigarettes
* Be able to read and speak English

Exclusion Criteria:

* Pregnant women
* Smokers who smoke exclusively roll-your-own cigarettes
* Smokers concurrently enrolled in another cessation study
* Smokers who smoke fewer than 7 cigarettes per week, on average
* Smokers who live in the same household as someone who has enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2149 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Quit attempts | Up to 4 weeks
  The primary outcome is a quit attempt during the 4 weeks of the study, reported at either 1, 2, 3, or 4 weeks. A quit attempt is defined as 24 hours without smoking.

SECONDARY OUTCOMES:
Change in quit intentions | 4 weeks
  Quit intentions will be measured at baseline pretest and posttest, 1, 2, 3, and 4 weeks using the 3-item quit intention scale developed by Klein, Zajac, and Monin (2009).
Successful Quitting | 4 weeks
  Successful quitting will be defined as self-reported smoking on 0 of the past 7 days at 4 weeks.
Change in forgoing a cigarette | 4 weeks
  Forgoing a cigarette will be measured at baseline pretest, 1, 2, 3, and 4 weeks as the frequency of butting out a cigarette or forgoing a cigarette in an effort to smoke less, using measures developed by the investigators.
Change in positive reinforcement attitudes | 4 weeks
  Positive reinforcement attitudes smoking attitudes will be measured at baseline pretest and posttest, 1, 2, 3, and 4 weeks using measures adapted from the Smoking Consequences Scale developed by Brandon & Baker (1991).
Change in negative reinforcement attitudes | 4 weeks
  Negative reinforcement attitudes will be measured at baseline pretest and posttest, 1, 2, 3, and 4 weeks using measures adapted from the Smoking Consequences Scale developed by Brandon & Baker (1991).
Change in perceived likelihood | 4 weeks
  Perceived likelihood of developing smoking-related health outcomes will be measured at baseline pretest, 2, and 4 weeks using measures developed by the investigators.
Change in frequency of conversations about warning labels | 4 weeks
  Frequency of conversations with other about the warning labels, health effects of smoking and quitting in the past week will be measured at baseline pretest, 1, 2, 3, and 4 weeks.
Fear | 4 weeks
  Fear will be measured at baseline posttest, 1, 2, 3, and 4 weeks using items developed by the investigators and adapted from Nonnemaker et al. (2010), Leshner et al. (2011), Watson et al. (1988), and Keller and Block (1996).
Cognitive elaboration | 4 weeks
  Cognitive elaboration will be measured at 1, 2, 3, and 4 weeks adapted from the Depth of Cognitive Processing Scale (Hammond, Fong, McDonald, Cameron, and Brown, 2003) and measures adapted from Fathelrahman et al (2010).

OTHER OUTCOMES:
Change in smoking quantity | 4 weeks
  Smoking quantity will be measured at baseline pretest, 1, 2, 3, and 4 weeks as the self-reported average number of cigarettes smoked per day during the past week. This measure is adapted from the Population Assessment of Tobacco and Health (PATH) Study (2013).
Change in cessation aid use | 4 weeks
  Use of cessation aids will be measured at baseline pretest, 1, 2, 3, and 4 weeks.
Change in e-cigarette use frequency | 4 weeks
  Frequency of e-cigarette use will be measured at 1, 2, 3, and 4 weeks as the number of days of use in the last 7 days. This measure is adapted from the Population Assessment of Tobacco and Health (PATH) Study (2013).
Initiation of e-cigarette use | 4 weeks
  Among never users of e-cigarettes at baseline pretest, initiation of e-cigarette use will be measured at 4 weeks.
Change in quit stage | 4 weeks
  Quit stage will be measured at baseline pretest and posttest, 1, 2, 3, and 4 weeks using a measure adapted from the International Tobacco Control (ITC) Policy Evaluation Survey.
Change in implementation intentions | 4 weeks
  Implementation intentions will be measured at baseline pretest and 4 weeks to assess how much participants have planned when to quit, how to quit, and how to deal with cravings after quitting.
Change in perceived severity | 4 weeks
  Perceived severity of developing various smoking-related health outcomes and of developing quitting side effects will be measured at baseline pretest, 2, and 4 weeks using measures adapted from Lyna (2002).
Change in anticipated regret | 4 weeks
  Anticipated regret of continuing to smoke and anticipated regret of quitting smoking will be measured at baseline pretest, 2, and 4 weeks using measures developed by the investigators.
Change in costs of quitting | 4 weeks
  Costs of quitting will be measured at baseline pretest, 1, 2, 3, and 4 weeks using measures adapted from McKee, O'Malley, Salovey, Krishnan-Sarin, and Mazure (2005).
Change in benefits of quitting | 4 weeks
  Benefits of quitting will be measured at baseline pretest, 1, 2, 3, and 4 weeks using measures adapted from McKee, O'Malley, Salovey, Krishnan-Sarin, and Mazure (2005).
Change in response efficacy | 4 weeks
  The response efficacy of quitting smoking will be measured at baseline pretest, 2, and 4 weeks using measures developed by the investigators.
Change in smoking cons | 4 weeks
  Cons of smoking will be measured at baseline pretest and posttest, 1, 2, 3, and 4 weeks using measures adapted from the Smoking Consequences Scale developed by Brandon & Baker (1991) and items from Velicer (1985).
Change in worry | 4 weeks
  Worry about the consequences of smoking will be measured at baseline pretest and posttest, 1, 2, 3, and 4 weeks using measures adapted from Dijkstra (2003), Ranby (2013) and Magnan (2009 and 2013).
Change in self-efficacy to quit smoking | 4 weeks
  Self-efficacy to quit smoking will be measured at baseline pretest, 2, and 4 weeks using measures adapted from Armitage (2007).
Change in pack attitudes | 4 weeks
  Pack attitudes will be measured at baseline pretest and 4 weeks using measures adapted from Moodie (2011).
Change in smoker prototypes | 4 weeks
  Positive and negative smoker prototypes will be measured at baseline pretest and posttest, 1, 2, 3, and 4 weeks using items developed by the investigators and adapted from the smoker prototype scale developed by McCool, Cameron, et al. (2010).
Change in e-cigarette user prototypes | 4 weeks
  Positive and negative e-cigarette user prototypes will be measured at baseline pretest and posttest, 1, 2, 3, and 4 weeks using items developed by the investigators and adapted from the smoker prototype scale developed by McCool, Cameron, et al. (2010).
Change in subjective norms | 4 weeks
  Subjective norms about smoking cessation will be measured at baseline pretest, 1, 2, 3, and 4 weeks using measures adapted from Armitage (2007) and Von Dras (2004).
Social reactions | 4 weeks
  Social reactions to the warning labels will be measured at baseline pretest, 1, 2, 3, and 4 weeks using measures developed by the the investigators to assess the nature, recipient and mode of communication about the warning labels, quitting smoking, and the health effects of smoking.
Perceived effectiveness | 4 weeks
  Perceived effectiveness of the warning labels will be measured at baseline post-test and 4 weeks using measures adapted from Hitchman, Driezen, Logel, Hammond, and Fong (2013), Trasher et al. (2012) & Cantrell et al (2013).
Avoidance | 4 weeks
  Avoidance of the warning label will be measured 1, 2, 3, and 4 weeks using measures adapted from the Population Assessment of Tobacco and Health Study (2014) and the Environics Research Group (2008), as well as measures developed by the investigators.
Reactance | 4 weeks
  Reactance to the warning label will be measured at baseline posttest, 1 and 4 weeks using a scale developed by the investigators.
Emotional reactions | 4 weeks
  Emotional reactions (i.e., anxiety, disgust, sadness, guilt, anger) will be measured at baseline posttest, 1, 2, 3, and 4 weeks using 12 items developed by the investigators and adapted from Nonnemaker et al. (2010), Leshner et al. (2011), Watson et al. (1988), and Keller and Block (1996).
Perceived understandability | 4 weeks
  Perceived understandability will be measured at baseline posttest and 4 weeks using a measure adapted from Cameron, Pepper, and Brewer (2013).
Attention/noticing | 4 weeks
  Attention/noticing of labels will be measured at baseline posttest, 1, 2, 3, and 4 weeks using measures adapted from Fathelrahman et al. (2010) and Nonnemaker et al. (2010).
Recall | 4 weeks
  Participants will be randomly assigned to be assessed unprompted recall of the image and text of their assigned warning label at 1, 2, 3 or 4 weeks.
Recognition | 4 weeks
  Participants will be randomly assigned to be assessed recognition of the image and text of their assigned warning label at either 1, 2, 3, or 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Brewer, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Prevention Research Center of the Pacific Institute for Research & Evaluation, Oakland, California
  - Pacific Institute for Research and Evaluation, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No
No patient level data will be shared with the general public or other researchers.

REFERENCES:
- [Derived] Brewer NT, Parada H, Hall MG, Boynton MH, Noar SM, Ribisl KM. Understanding Why Pictorial Cigarette Pack Warnings Increase Quit Attempts. Ann Behav Med. 2019 Mar 1;53(3):232-243. doi: 10.1093/abm/kay032. PMID 29850764
- [Derived] Parada H Jr, Hall MG, Boynton MH, Brewer NT. Trajectories of Responses to Pictorial Cigarette Pack Warnings. Nicotine Tob Res. 2018 Jun 7;20(7):876-881. doi: 10.1093/ntr/ntx182. PMID 29059340
- [Derived] Brewer NT, Hall MG, Noar SM, Parada H, Stein-Seroussi A, Bach LE, Hanley S, Ribisl KM. Effect of Pictorial Cigarette Pack Warnings on Changes in Smoking Behavior: A Randomized Clinical Trial. JAMA Intern Med. 2016 Jul 1;176(7):905-12. doi: 10.1001/jamainternmed.2016.2621. PMID 27273839
- [Derived] Brewer NT, Hall MG, Lee JG, Peebles K, Noar SM, Ribisl KM. Testing warning messages on smokers' cigarette packages: a standardised protocol. Tob Control. 2016 Mar;25(2):153-9. doi: 10.1136/tobaccocontrol-2014-051661. Epub 2015 Jan 6. PMID 25564282